CLINICAL TRIAL: NCT03873610
Title: Resiliency Training in Adolescents With NF1 and NF2; A Randomized Controlled Trial Via Secure Live Video Conferencing to Improve Emotional, Social and Physical Function
Brief Title: Resiliency Training in Adolescents With NF1 and NF2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019P000625
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromatoses
MeSH Terms: conditions — Neurofibromatoses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress and Symptom Management Program 1 (Experimental)
  Interventions: Behavioral: Stress and Symptom Management Program 1
- Stress and Symptom Management 2 (Experimental)
  Interventions: Behavioral: Stress and Symptom Management Program 2

INTERVENTIONS:
Behavioral: Stress and Symptom Management Program 1 — The Stress and Symptom Management Program 1 introduces and reinforces stress and symptom management for adolescents with NF. The program consists of 8 weekly 45 minute sessions, delivered through videoconferencing.
  Arms: Stress and Symptom Management Program 1
Behavioral: Stress and Symptom Management Program 2 — The Stress and Symptom Management Program 2 introduces and reinforces stress and symptom management for adolescents with NF. The program consists of 8 weekly 45 minute sessions, delivered through videoconferencing.
  Arms: Stress and Symptom Management 2

SUMMARY:
This randomized controlled trial for resiliency training in adolescents with Neurofibromatosis 1 and Neurofibromatosis 2 via secure live video to determine the efficacy two stress and symptom management programs. Both programs are 8 week group programs.

DETAILED DESCRIPTION:
Neurofibromatosis (NFs) are rare genetic conditions with cure. Adolescents with NF experience more symptoms of depression and anxiety, higher levels of stress associated with coping with NF symptoms, lower levels of self esteem, difficulties with social skills and social support, high rates of learning disabilities, and more pain as compared with the general population norms.

The aims of this study are to compare the effect of two stress and symptom management programs tailored for adolescents with neurofibromatosis on quality of life and psychosocial functioning. We will also examine the degree to which treatment-dependent improvements in quality of life are mediated by improvements in depression, pain intensity and pain interference.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of NF1 or NF2 and is between the ages of 12-17
* Is capable of completing and fully understanding the informed consent process/assent and the study procedures and assessments in English; has parental approval for participation
* English speaking and at least a 3rd grade self-reported and parent reported reading level
* Self reported/parent reported difficulties coping with stress and NF symptoms

Exclusion Criteria:

* Has major medical co-morbidity not NF related expected to worsen in the next 12 months
* Recent (within past 3 months) change in antidepressant medication
* Recent participation in cognitive behavioral therapy or relaxation therapy (within past 3 months)
* Has significant mental health diagnosis requiring immediate treatment (e.g., untreated bipolar disorder, psychotic disorder, active substance dependence)
* Unable or unwilling to complete assessments electronically via REDCap
* Unable or unwilling to participate in group videoconferencing sessions
* Unable or unwilling to participate along with at least 1 parent in a video screening session

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Health Quality of Life | 0 weeks, 8 weeks, 6 months,12 months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; Higher score indicates higher QoL
Change in Psychological Health Quality of Life | 0 weeks, 8 weeks, 6 months,12 months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; Higher score indicates higher QoL

SECONDARY OUTCOMES:
Social relationships Quality of Life | 0 weeks, 8 weeks, 6 months,12 months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; Higher score indicates higher QoL
Environmental Quality of Life | 0 weeks, 8 weeks, 6 months, 12 months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; Higher score indicates higher QoL
Depression | 0 weeks, 8 weeks, 6 months, 12 months
  Patient Health Questionnaire (PHQ-9) Adolescent Version; 0-27; Higher score indicates more symptoms of depression
Anxiety | 0 weeks, 8 weeks, 6 months, 12 months
  Generalized Anxiety Disorder (GAD-7) Questionnaire; 0-21; Higher score indicates more symptoms of anxiety
Pain intensity | 0 weeks, 8 weeks, 6 months, 12 months
  Numerical Rating Scale; 0-10; Higher score indicates more intense pain.
Pain interference | 0 weeks, 8 weeks, 6 months, 12 months
  Pain Interference Index (PII); 0-36; Higher score indicates more pain interference

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No